CLINICAL TRIAL: NCT01447641
Title: Characterisation of Sleep and Circadian Physiology in Individuals With Cluster Headache
Brief Title: Sleep, Circadian Rhythms and Cluster Headache
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CRC301
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cluster Headache
Keywords: Cluster Headache; Trigeminal Autonomic Cephalalgias; Sleep; Circadian Rhythms
MeSH Terms: conditions — Cluster Headache; Trigeminal Autonomic Cephalalgias | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood hormonal and circulating lymphocyte mRNA assays
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cluster headache: Cluster headache sufferers (both chronic and episodic)
  Interventions: Other: Polysomnography; Other: Actigraphy

INTERVENTIONS:
Other: Polysomnography — Overnight physiological recording of sleep
Other: Actigraphy — Wristwatch activity to measure basic rest activity cycle and sleep efficiency

SUMMARY:
The purpose of this study is to assess both the sleep and circadian (24-hourly biological rhythms) physiology of people with cluster headache. For sufferers with the episodic form of the disorder this will involve observation at two separate time points, once when experiencing attacks (in-bout) and once when attack free (out-of-bout).

The study will include measurement of basic rest-activity patterns, sleep timing and timing of individual attacks, as well as a more detailed study recording sleep and circadian rhythms under clinical conditions over consecutive nights.

Studying the differences in these processes in single individuals when they are both experiencing and free from attacks might provide insight into the brain mechanisms involved in triggering the bouts of attacks and individual attacks themselves. An improved understanding of this area may help design improved treatment options in future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cluster headache or closely related primary headache disorder

Exclusion Criteria:

* Abnormality on screening investigations that increase risk of participation
* Alcohol consumption exceeding 21 units per week

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cluster headache sufferers (both of the episodic and chronic cluster headache) Related headache disorders
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
amplitude and phase of circadian rhythm of melatonin | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Nesbitt, BM BCh MRCP, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, University of Surrey, Guildford, United Kingdom